CLINICAL TRIAL: NCT05789706
Title: Use of a Smart-phone Based Medication Adherence Platform to Improve Outcomes in Uncontrolled Non-insulin Dependent Diabetes Among Veterans: a Pragmatic, Point-of-care, Implementation Effectiveness Pilot Study
Brief Title: Use of a Smart-phone Based Medication Adherence Platform to Improve Outcomes in Uncontrolled Non-insulin Dependent Diabetes Among Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Sierra Nevada Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Amneet Rai, Associate Chief of Pharmacy - Health Outcomes and Analytics, VA Sierra Nevada Health Care System
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1655381
Record Dates: First submitted 2022-10-24; First posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Diabetes; Diabete Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This study will employ a case-crossover design where patients will undergo both a standard of care arm as well as an intervention arm. Half of the study participants will be randomized and enrolled in the standard of care arm for the initial 3 months and then transition to the intervention arm for 3 months. The remaining patients will be enrolled in the intervention arm for the initial 3 months and then transitioned to the standard of care arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Patients will have Dayamed Arthur a novel intelligent medication adherence platform installed on their smartphone and configured with their pharmacy data providing accurate prompts and reminders to patients to take medications as directed In addition to the prompts patient all auditable information will be relayed to their PACT CPS through a provider dashboard allowing for timely and directed clinical intervention. Dayamed Arthur will provide automated alerts to the patients care team in specific scenarios.
  Interventions: Behavioral: Dayamed Arthur a novel intelligent medication adherence platform
- Standard of Care Arm (No Intervention): Study subjects will be counseled on medication adherence and strategies to remember how to take their medications correctly. Study subjects will then be followed as clinically indicated by their clinical care team.

INTERVENTIONS:
Behavioral: Dayamed Arthur a novel intelligent medication adherence platform — Novel smart phone adherence application configured with subject pharmacy data providing accurate reminders of when to take medications and providing auditable user feed back to clinical care teams for patient response directed provider intervention.
  Arms: Intervention Arm

SUMMARY:
The purpose of this study is to determine if a novel smartphone-based medication adherence platform accompanied by directed pharmacist intervention can improve A1c control and medication compliance in non-insulin dependent diabetics.

DETAILED DESCRIPTION:
This study will employ a case-crossover design where patients will undergo both a standard of care arm as well as an intervention arm (See Figure 1). Half of the study participants will be randomized and enrolled in the standard of care arm for the initial 3 months and then transition to the intervention arm for 3 months. The remaining patients will be enrolled in the intervention arm for the initial 3 months and then transitioned to the standard of care arm.

Primary outcomes will be the change from pre-intervention baseline in hemoblobin A1c (HgA1c) between the Dayamed Arthur platform and standard of care.

Secondary outcomes will include change in MAS, the change in RMA from week 1 of intervention arm to week 12, comparison of historical MPR and PDC with patient's RMA at week 1 of intervention arm, and correlation of change in RMA and MAS score during intervention arm. Furthermore, we will measure sustained change in MAS in the patient population who begin study in the intervention arm and are subsequently transitioned to standard of care. We will also collect information patient usability/acceptability and provider satisfaction with the Dayamed Arthur platform.

Exploratory outcomes will include potential reduction in healthcare resource utilization based on avoidance of therapy escalation in patients with improved compliance, as well as psychosocial factors associated with improved adherence

Reduction of HgbA1c by 0.5% from pre-intervention baseline for individuals on the DayaMed intervention compared to standard of care

ELIGIBILITY:
Inclusion Criteria:

* Assigned primary care provider at VA Sierra Nevada Healthcare System (VASNHCS)
* Diagnosis of type 2 diabetes
* Own a smart phone/tablet
* HgbA1c drawn at or within 30 days of study enrollment.
* Uncontrolled A1c defined as an A1c >9 in the following order of preference

  * Last 3 A1cs >9% in the last 2 year
  * Last 2 A1cs >9% in the last 2 years
  * Last A1c >9% in the last 2 years
  * 2-year average A1c >9%

Exclusion Criteria:

* Actively on insulin therapy
* Unable to install DayaMed application onto their phone/tablet
* Unable to load medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Change from pre-intervention baseline in hemoblobin A1c | 3 months
  The change from pre-intervention baseline in hemoblobin A1c (HgA1c) to 3 months in the intervention arm compared to change from baseline to 3 months in the standard of care arm

SECONDARY OUTCOMES:
Change in Medication Adherence Score from baseline | 3 months
  change from baseline to 3 months in medication adherence score in the intervention arm compared to change from baseline to 3 months in medication adherence score in the standard of care arm

CONTACTS AND LOCATIONS:
Locations (1):
- VA Sierra Nevada Health Care System, Reno, Nevada, United States

IPD SHARING:
Plan to Share IPD: No